CLINICAL TRIAL: NCT02176096
Title: Comparison of the Effect of a Novel Starch (Glycosade) Versus Gastrostomy Tube-Dextrose Infusion on Overnight Euglycaemia Control in Children With Glycogen Storage Disease Type I: Open Label Demonstration Trial
Acronym: Glycosade GSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Co-Investigator - Dr. Cheryl Rockman-Greenberg (Unknown)
Responsible Party: Principal Investigator, Dr. Aizeddin (Aziz) Mhanni, Associate Professor, Department of Pediatrics and Child Health, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2013-097
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Glycogen Storage Disorder Type 1; Hypoglycemia; Cornstarch; Glycosade
MeSH Terms: conditions — Hypoglycemia | interventions — octenyl succinic anhydride-modified starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glycosade (Experimental)
  Interventions: Dietary Supplement: Glycosade

INTERVENTIONS:
Dietary Supplement: Glycosade
  Other Names: Modified starch

SUMMARY:
The objective of this demonstration project is to compare a novel long-acting starch, Glycosade, a hydrothermally processed high amylopectin maize starch, versus gastrostomy tube-dextrose infusion in maintaining euglycaemia overnight in children with GSD-I. Glycosade has been reported to increase the duration of euglycaemia. Its slow release and longer periods of normal blood sugar achieved would preclude the need for the overnight dextrose infusion and eliminate the need for the surgical insertion of a gastrostomy tube for this purpose. Glycosade also reportedly causes fewer gastrointestinal side effects, thus potentially improving compliance to therapy. The investigators intend to evaluate Glycosade in our patients and determine its efficacy on glucose control, on the length of normoglycemia achieved and to determine if there are reduced side effects in our patients with GSD-I. This will be accomplished by an open label study of Glycosade in GSD-I patients who consent to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GSD Type 1
* Age >5 years

Exclusion Criteria:

* n/a

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Normal Blood Glucose | Overnight
  With the use of Glycosade blood glucose would be maintained for 8 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Chrildren's Hospital Research Institute of Manitoba, Winnipeg, Manitoba, Canada